CLINICAL TRIAL: NCT05122533
Title: Reliability Study of the Clinical Limb-length Measurements Methods Applied in Healthy Volunteers
Brief Title: Reliability of Clinical Limb-length Measurements Methods
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: UP-CC-Ortho-LimbLength
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Leg Length Inequality
Keywords: leg length inequality; leg length discrepancy; EOS 2D/3D; physical examination; length measurement
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: 18-30 year-old, healthy volunteers
  * Age: 18-30 years
  * BMI: <30
  * No previous surgery on lower limb or spine
  * No known developmental disorder
  * Without any orthopaedic complaint
  Interventions: Diagnostic Test: EOS; Diagnostic Test: Clinical limb length measurements

INTERVENTIONS:
Diagnostic Test: EOS — EOS Micro Dose imaging will be done. SterEOS lower limb alignment reconstruction will be performed measuring the lim length.
  Other Names: EOS 2D/3D scanning and SterEOS 3D reconstruction
Diagnostic Test: Clinical limb length measurements — Clinical measurement of both lower limbs' length, 3 times in 3 different days by 3 observers.
  * bony markers position (heel contour, patella and medial malleolus) in resupinate and side position also
  * tape measuring:
    * Spina iliaca anterior superior - medial malleolus
    * umbilicus - medial malleolus
    * greater trochanter - lateral malleolus
    * in standing, sitting, resupinate and side position

SUMMARY:
There are numerous ways to measure limb length discrepancy in the clinical practice, although their reliability and accuracy are not well known. In our prospective diagnostic study we aimed to test the most popular methods and compare their results to EOS 3D reconstructions data.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-30 years
* BMI: < 30
* Without orthopaedic complaint

Exclusion Criteria:

* Previous surgery on lower limb or spine
* Developmental disorder in the patients history

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young, healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Radiological limb length | 6 months
  Limb length based on SterEOS 3D measurement
Intra- and interobserver reliability of the clinical lower limb measurements methods | 6 months
  Intra- and interobserver reliability of clinical length measuring methods will be calculated using the 3 separated measurement of the 3 observers.
Accuracy of the clinical lower limb measurements methods | 6 months
  Comparing the results of the radiological and clinical limb length results using the third measurement of the observers.

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Schlegl, MD, PhD, Study Chair — University of Pecs Medical School, Department of Orthopaedics
Locations (1):
- Universtify of Pecs, Department of Orthopaedics, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No